CLINICAL TRIAL: NCT04826445
Title: USE OF 18FDG PET-CT TO PREDICT THE RESPONSE OF MANDIBULAR OSTEORADIONECROSIS TO THE PENTOCLO PROTOCOL WITH DOCUMENTED ANTIBIOTHERAPY
Acronym: PENTOTEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00965-52; 2019/2931 (Other: CSET number)
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Mandibular Osteoradionecrosis
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included in PENTOCLO protocol: We perform a prospective study with inclusions of all consecutive patients with osteoradionecrosis eligible for PENTOCLO.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Imaging collection

SUMMARY:
This study is created in order to refine and reduce the duration between the medical and surgical therapeutic sequences (when the surgery is necessary) in these fragile patients knowing that conventional radiological changes can only be observed with a delay comprised between 3 and 6 months starting from observed clinical changes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic osteoradionecrosis with a PENTOCLO protocol indication (decided in a multi-disciplinary staff).
2. Patient should understand to any protocol-specific procedures performed. Patient who did not object to participate after being informed of the study. Patient should be able and willing to comply with study visits and procedures as per protocol.
3. Patients must be affiliated to a social security system or beneficiary of the same.
4. Patients must be over 18 years old (legal age).

Exclusion Criteria:

1. Excluded forms of the disease: mandibular osteoradionecrosis complicated by mandibular fracture and / or hyperalgesic (resistant to analgesic treatment of stage III).
2. Contraindications specific to the treatment under study (allergy to one of the PENTOCLO treatments, contraindication to 18FDG PET-CT).
3. Associated pathology that contra-indicate on of the PENTOCLO treatment.
4. Pregnant woman, declaring likely to be pregnant or breastfeeding. Chilbearing age women must declare not being pregnant and use effective contraception.
5. Impossibility to submit to the medical follow-up of the test for geographical, social or psychological reasons.
6. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or unable to express its opposition to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mandibular osteoradionecrosis treated in the PENTOCLO protocol
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
diagnosis performance of 18-FDG PET-CT | up to 3 months
  Evaluate the diagnosis performance of 18-FDG PET-CT with the criteria of Mandibular mean FDG uptake compared between the reference test and at 3 months: ΔSUVmean

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: Undecided